CLINICAL TRIAL: NCT04625868
Title: Effectiveness of a Preoperative Educational Video for Reducing Opioid Consumption After Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Principal Investigator, David Kalainov, Clinical Professor of Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00211034
Record Dates: First submitted 2020-07-03; First posted 2020-11-12 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Opioid Use; Hand Injuries and Disorders; Surgery
MeSH Terms: conditions — Hand Injuries; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soft tissue surgery - preoperative video (Experimental): Patients > 18 years old undergoing elective hand surgery (soft tissue) for which the surgeon is planning to prescribe opioids for postoperative pain control.
  Interventions: Other: Educational video
- Soft tissue surgery - no video (No Intervention): Patients > 18 years old undergoing elective hand surgery (soft tissue) for which the surgeon is planning to prescribe opioids for postoperative pain control.
- Bone/joint surgery - preoperative video (Experimental): Patients > 18 years old undergoing elective hand surgery (bone/joint) for which the surgeon is planning to prescribe opioids for postoperative pain control.
  Interventions: Other: Educational video
- Bone/joint surgery - no video (No Intervention): Patients > 18 years old undergoing elective hand surgery (bone/joint) for which the surgeon is planning to prescribe opioids for postoperative pain control.

INTERVENTIONS:
Other: Educational video — Patients will watch a preoperative educational video on proper opioid use and disposal.
  Arms: Bone/joint surgery - preoperative video; Soft tissue surgery - preoperative video

SUMMARY:
This study seeks to determine if watching a preoperative educational video influences opioid consumption and proper disposal following elective hand surgery.

DETAILED DESCRIPTION:
This study seeks to determine if watching a preoperative educational video influences opioid consumption and proper disposal following elective hand surgery. Patients undergoing elective hand surgery are randomized to either watch a preoperative educational video or not. Patients are asked to record their pain medication usage postoperatively, as well as their daily pain levels and satisfaction with their pain control after surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective hand surgery
* surgeon is planning to prescribe opioids for postoperative pain control

Exclusion Criteria:

* emergent surgery
* surgeon not planning to prescribe opioids for postoperative pain control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Morphine milliequivalents consumed in 2 weeks postoperatively | 2 weeks after surgery
  Total morphine mEq consumed in 2 weeks after surgery

SECONDARY OUTCOMES:
Visual Analog Scale | 2 weeks after surgery
  Average daily Visual Analog Scaled pain score recorded after surgery. Pain will be recorded on a scale from 0 (no pain) to 10 (worst pain possible).
Patient satisfaction | 7-10 days after surgery
  Patient satisfaction with pain control after surgery. Satisfaction will be measured on a Likert scale with the following question: "How satisfied have you been with your pain management after surgery?". Answer choices are: Very unsatisfied, unsatisfied, neutral, satisfied, very satisfied.
Proper disposal | 2 weeks after surgery
  Self-reported proper disposal of unused opioids after surgery. Patients will be asked in a postoperative survey if they used all of the pills in their initial postoperative prescription. If they did not, they will be asked "Have you disposed of your unused opioids via a DEA-approved method (I.e. at a pharmacy or other safe location?)" as a yes or no question.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Kalainov, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No